CLINICAL TRIAL: NCT06635928
Title: Assessing Fatigue and Attention in Myalgic Encephalomyelitis/Chronic Fatigue Syndrome Patients Before and After Treatment With Bright Light Therapy: a Prospective Randomized Controlled Crossover Study
Brief Title: Bright Light Therapy in ME/CFS Patients
Acronym: BLTME
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of Vienna (Other)
Responsible Party: Principal Investigator, Stefan Seidel, Professor, Medical University of Vienna
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: MUVienna
Record Dates: First submitted 2024-10-07; First posted 2024-10-10 (Actual); Last update posted 2024-10-10 (Actual); Status verified 2024-10

CONDITIONS: Myalgic Encephalomyelitis/Chronic Fatigue Syndrome
Keywords: bright light therapy; ME/CFS; attention testing; fatigue
MeSH Terms: conditions — Fatigue Syndrome, Chronic; Fatigue | interventions — Ultraviolet Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Wait list (No Intervention)
- Intervention (Experimental): Bright light therapy for 2 weeks, 30min a day
  Interventions: Device: Bright light therapy

INTERVENTIONS:
Device: Bright light therapy — 30min daily of 10.000 lux bright light therapy
  Arms: Intervention

SUMMARY:
In this study patients with Myalgic Encephalomyelitis/Chronic Fatigue Syndrome (ME/CFS) will receive bright light therapy through portable lamps for 2 weeks. They will either start with this treatment and then go through a wash-out period of two weeks followed by a wait period of two weeks or they will start with the wait period, followed by a wash-out period, followed by the treatment phase. Patients are asked to fill out questionnaires (rating their level of fatigue) and they go through a standardized computer test assessing their attention levels, both at multiple times throughout the study. The aim of this study is to find out if treatment with bright light will improve subjective fatigue levels and objective attention levels inME/CFS patients.

DETAILED DESCRIPTION:
Chronic Fatigue Syndrome (CFS), also referred to as Myalgic Encephalomyelitis (ME), is a chronic, debilitating condition of unknown etiology. Bright light therapy (BLT) has shown promising results in studies investigating its effect in patients with neurological disorders experiencing fatigue symptoms (Mateen et al., 2020, Sinclair et al., 2014, West et al., 2019). Since effective and low to no side effect therapies are duly needed for the treatment of ME/CFS, we propose a randomized-controlled treatment approach with bright light therapy (BLT).

In this proposed study, a total of 38 out-patients with a diagnosis of ME/CFS according to the criteria of the Institute of Medicine will be randomly assigned to a crossover design starting out either with BLT or being waitlisted for the course of two weeks. Portable light boxes emitting full-spectrum visible light with a luminance intensity of 10,000 lux measured at a distance of 50 cm will be used at the participants' home for 2 weeks.

Primary outcome of the study will be the level of fatigue before and after treatment as operationalized by the Chalder Fatigue Score. Secondary outcomes include the objective activity pattern as measured by actigraphy as well as cognitive and metacognitive functioning assessed before and after treatment.

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of ME/CFS according to the IOM (IOM, 2015)
* Chalder Fatigue Score of ≥ 18 points (Likert scoring)
* age 18-60 years;
* ability to give informed consent.

Exclusion Criteria:

* Comorbidities explaining current fatigue symptoms such as sleep-wake disorders (narcolepsy, sleep apnea, periodic limb movements during sleep and irregular sleep-wake-rhythm), untreated hypothyroidism and iatrogenic conditions such as side effects of medication.
* Previous treatment with BLT (> 10.000 lux) for a duration of >2 weeks.
* Previously diagnosed medical conditions such as malignancies and hepatitis B or C virus infection.
* Any past or current diagnosis of bipolar affective disorder; schizophrenia; dementias of any subtype; anorexia nervosa; or bulimia nervosa.
* Alcohol or other substance abuse disorders within 2 years before the onset of the chronic fatigue and at any time afterward.
* Severe obesity as defined by a body mass index equal to or greater than 45.
* Medication use interacting with the circadian rhythm such as regular intake of sleeping pills, sleep-inducing antidepressant medication, and immunosuppressive medication.
* >20 points in the HDRS-17
* >10 points in GAD-7 in the psychiatric screening process
* Pregnancy
* Change in regimen of ongoing treatment with antidepressants or stimulants within 4 weeks before study inclusion

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 36 (Actual)
Dates: Start 2021-01-01 (Actual); Primary Completion 2024-03-25 (Actual); Study Completion 2024-03-25 (Actual)

PRIMARY OUTCOMES:
Chalder Fatigue Score | As a baseline variable: day 1 of inclusion in the study, day 7 before treatment/wait list, day 21 after treatment/wait list, day 35 before treatment/wait list and day 42 after treatment/wait list
  subjective Fatigue score

SECONDARY OUTCOMES:
Test of Attentional Performance | On day 7 before treatment/wait list, day 21 after treatment/wait list, day 35 before treatment/wait list and day 42 after treatment/wait list
  three subtests of attention

CONTACTS AND LOCATIONS:
Locations (1):
- Medical University of Vienna, Vienna, Austria

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Ludwig B, Hauer L, Bock M, Schillerwein-Kral C, Weyer L, Moser D, Zehetmayer S, Trimmel K, Seidel S. Assessing fatigue in myalgic encephalomyelitis/chronic fatigue syndrome patients before and after treatment with bright light therapy: A prospective randomized controlled crossover study. Sleep Med. 2025 May;129:369-374. doi: 10.1016/j.sleep.2025.03.003. Epub 2025 Mar 14. PMID 40120538